CLINICAL TRIAL: NCT00727740
Title: A Prospective, Multicenter, Randomized, Double-blind Controlled Study to Determine Whether a Single Dose of Intraduodenal Indomethacin Can Decrease the Incidence and Severity of Post-ERCP Pancreatitis
Brief Title: A Double-blind Study to Determine if Intraduodenal Indomethacin Can Decrease the Incidence of Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0502027420
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatitis
Keywords: Cholangiopancreatography, Endoscopic Retrograde; Pancreatitis; Indomethacin
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Indomethacin liquid suspension 100 mg (25 mg/5ml) which is 20 cc of suspension instilled via a Teflon catheter (the end of which is passed through the biopsy channel of the endoscope) and situated into the duodenum. Following instillation of the suspension, the catheter is flushed with 5 cc of normal saline.
  Interventions: Drug: Indomethacin
- 2 (Placebo Comparator): Placebo suspension in the same volume (20 cc) which is instilled via a Teflon catheter (the end of which is passed through the biopsy channel of the endoscope) and situated into the duodenum. The placebo suspension is also flushed with 5 cc of normal saline.
  Interventions: Drug: Placebo suspension

INTERVENTIONS:
Drug: Indomethacin — Indomethacin 100 mg liquid suspension (25 mg/5 ml) which is 20 cc of suspension is instilled via a Teflon catheter (the end of which is passed through the biopsy channel of the endoscope) and situated into the duodenum. Following instillation of the suspension, the catheter is flushed with 5 cc of normal saline.
  Arms: 1
Drug: Placebo suspension — A placebo suspension which is made by the Investigational Drug Service (IDS) by adding the appropriate dye coloring to normal saline so that the appearance is identical to the indomethacin suspension. The placebo solution is also instilled via a Teflon catheter (the end of which is passed through the biopsy channel of the endoscope) and situated into the duodenum. Following instillation of the placebo suspension, the catheter is flushed with 5 cc of normal saline.
  Arms: 2

SUMMARY:
The purpose of this research study is to determine if indomethacin, an anti-inflammatory medication in a class of medications known at NSAIDs (non-steroidal anti-inflammatory drugs) can reduce the risk of pancreatitis after Endoscopic Retrograde Cholangio-Pancreatography (ERCP.) The hypothesis is that indomethacin decreases the incidence and severity of post-ERCP pancreatitis. Patients who are scheduled to undergo a ERCP will be enrolled. Following ERCP, patients will be randomized to receive a dose of indomethacin or placebo (an inactive substance) instilled into the duodenum via the biopsy channel of the duodenoscope. All patients will be observed for 4 hours following ERCP which is part of routine clinical practice. Patients with minimal pain will be discharged after this 4 hour observation period. All patients will have baseline serum amylase levels which are repeated 2 to 4 hours after the ERCP has been completed. Patients who have significant abdominal pain will be hospitalized and evaluated for pancreatitis. Patients discharged to home will be contacted by telephone the following day to ask them if they have had any complications of ERCP.

DETAILED DESCRIPTION:
Post-ERCP pancreatitis is likely due to the patient's inflammatory response to duct instrumentation during the procedure and severity is based on the magnitude of this response. Phospholipase A2 (PLA2) plays a pivotal role in inflammation since it regulates many pro-inflammatory mediators, including prostaglandins, leukotrienes, and platelet activating factor. NSAIDs inhibit PLA2, and indomethacin is the most potent clinically available PLA2 inhibitor. Our study hypothesis is that treatment with indomethacin will reduce the inflammatory response to ERCP, and therefore lessen the incidence and severity of post-ERCP pancreatitis.

Aim: We plan to conduct a prospective, multicenter, randomized, placebo-controlled trial to determine if a single dose of 100 mg indomethacin suspension instilled into the duodenum by the endoscope immediately following ERCP can reduce the incidence and severity of post-ERCP pancreatitis.

Patients scheduled to undergo diagnostic or therapeutic ERCP would be serially enrolled. Standard indications for ERCP will include the following: evaluation of obstructive jaundice, unexplained pancreatitis, recurrent pancreaticobiliary pain and abnormal liver tests. Those patients who are deemed to be at increased risk of pancreatitis (suspected sphincter of oddi dysfunction, age < 40 yrs, normal bilirubin, prior post ERCP pancreatitis, difficult cannulation, pancreatic duct injection, pancreatic duct sphincterotomy, undergoing pre-cut sphincterotomy and balloon dilation of the biliary sphincter) would undergo placement of a 3 French pancreatic stent at the time of ERCP. Prospective randomized studies have demonstrated a marked decrease in post-ERCP pancreatitis rates in high risk patients who have undergone pancreatic stenting. Following ERCP and therapy (if required), they would be randomized to receive a dose of indomethacin or placebo instilled into the duodenum via the biopsy channel of the duodenoscope. Patients as well as physicians and nurses performing the procedure and overseeing the study will be unaware of treatment assignments.

All of the endoscopic and clinical practices will follow the current standard of care of the Yale interventional endoscopy department. Participation in the study will not alter this in any way. The experimental intervention is limited to the administration of a single dose of indomethacin, injected into the endoscope channel prior to removal of the scope at the conclusion of the ERCP and subsequent monitoring for signs and symptoms of post-ERCP pancreatitis, much of which is also part of routine clinical practice.

At the end of the procedure the details of the endoscopic maneuver are recorded, including ease/difficulty of cannulation, sphincterotomy (biliary and/or pancreatic) performed, number of cannulations, number of pancreatic duct injections, technique of sphincterotomy (Needle Knife/Stent vs pull-type) and duct diameters.

All patients will be observed for 4 hours following ERCP which is part of the routine clinical practice following ERCP. Patients with minimal pain will be discharged after a 4-hour period of observation. All patients will have baseline serum amylase levels which will be repeated 4 hours after the ERCP has been completed. Patients with significant abdominal pain following ERCP will be hospitalized overnight and evaluated for post-ERCP pancreatitis with monitoring of vital signs, urinary output and serum amylase levels the following morning. Patients with ongoing symptoms at 48 hours and later will undergo imaging with either abdominal ultrasonography or CT scanning. This also represents current standard clinical practice.

Patients discharged home will be contacted by telephone the following day to assess for complications including post-ERCP pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ERCP as part of their clinical care.

Exclusion Criteria:

* Pancreatitis within 60 days of ERCP
* Age less than 18 years
* Pregnant patients
* Patients who have received NSAIDs within the past 7 days
* Patients with a previous allergy to NSAIDs
* Patients who were previously enrolled in the study
* Patients with a history of peptic ulcers, gastrointestinal bleeding, on anticoagulants and/or with a bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2005-08; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Jamidar, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1- Indomethacin: Indomethacin liquid suspension 100 mg (25 mg/5ml) which is 20 cc of suspension instilled via a Teflon catheter (the end of which is passed through the biopsy channel of the endoscope) and situated into the duodenum. Following instillation of the suspension, the catheter is flushed with 5 cc of normal saline.
  Indomethacin: Indomethacin 100 mg liquid suspension (25 mg/5 ml) which is 20 cc of suspension is instilled via a Teflon catheter (the end of which is passed through the biopsy channel of the endoscope) and situated into the duodenum. Following instillation of the suspension, the catheter is flushed with 5 cc of normal saline.
- 2- Placebo: Placebo suspension in the same volume (20 cc) which is instilled via a Teflon catheter (the end of which is passed through the biopsy channel of the endoscope) and situated into the duodenum. The placebo suspension is also flushed with 5 cc of normal saline.
  Placebo suspension: A placebo suspension which is made by the Investigational Drug Service (IDS) by adding the appropriate dye coloring to normal saline so that the appearance is identical to the indomethacin suspension. The placebo solution is also instilled via a Teflon catheter (the end of which is passed through the biopsy channel of the endoscope) and situated into the duodenum. Following instillation of the placebo suspension, the catheter is flushed with 5 cc of normal saline.
Period: Overall Study
Arm/Group | 1- Indomethacin | 2- Placebo
Started | 56 | 61
Completed | 56 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- Indomethacin | 2- Placebo | Total
Number analyzed (Participants) | 56 | 61 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (18.3) | 56.6 (13.5) | 55.4 (16.1)
Gender [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Pancreatitis Rate
Description: Pancreatitis was operationally defined as post-ERCP pancreatitis (PEP). PEP was defined as abdominal pain with elevated serum amylase level (3 times above the upper limit of normal). The change in Pancreatitis rate calculated as the percentage of participants with pancreatitis at baseline minus percentage of participants with pancreatitis at 24 hours.
Time Frame: 24 hours
Measure: Number; unit: percentage of participants with PEP
Arm/Group | 1- Indomethacin | 2- Placebo
Number analyzed (Participants) | 56 | 61
percentage of participants with PEP | 16.1 | 4.9

ADVERSE EVENTS:
Arm/Group | 1- Indomethacin | 2- Placebo
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/61
Other Adverse Events (participants affected / at risk) | 0/56 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes